CLINICAL TRIAL: NCT01919775
Title: Basal Forebrain Amnesia After Surgery for Anterior Communicating Aneurysm： High Resolution 3-dimensional (3D) Magnetic Resonance (MR) Imaging Findings
Brief Title: Amnesia After Surgery for Anterior Communicating Aneurysm： High Resolution Magnetic Resonance (MR) Imaging Findings
Status: Completed | Type: Observational
Sponsor: Tohoku University (Other)
Responsible Party: Principal Investigator, Shunji MUGIKURA, Principal Investigator, Associate professor of Departmetn of Diagnostic radiology, Tohoku University
Other Study IDs: tohoku-ACoA amnesia MRI
Record Dates: First submitted 2013-08-07; First posted 2013-08-09 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Subarachnoid Hemorrhage; Cerebral Aneurysm; Amnesia
MeSH Terms: conditions — Subarachnoid Hemorrhage; Intracranial Aneurysm; Amnesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
To clarify whether amnesia after treatment of anterior communicating aneurysm (ACoA)is related to infarcts caused by occlusion or damage of the perforating artery of the ACoA, we used 3.0-T 3D high resolution MR imaging to identify and localize infarcts in patients with amnesia following treatment of ACoA aneurysm.

DETAILED DESCRIPTION:
Cohort register is made by experienced neuropsychologists in our institute.

MR imaging and data storage is in the department of diagnostic radiology of our institute.

MR images are evaluated by two neuroradiologists using a work station.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Amnesia

Exclusion Criteria:

Severe decreased intellectual function

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with amnesia following surgical treatment of the ACoA aneurysm.
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2007-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
cerebral infarction identified and localized in the basal forebrain on MR imaging | within 15 months from the aneurysmal treatment(an expected average 4 months)

CONTACTS AND LOCATIONS:
Overall Officials: Shoki Takahashi, Professor, Study Director — Department of Diagnostic Radiology, Tohoku University, Graduate School of Medicine, Sendai, Japan